CLINICAL TRIAL: NCT07217873
Title: IntraVenous Iron in Kids With Iron Deficiency and Scoliosis
Brief Title: IntraVenous Iron in Kids With Iron Deficiency and Scoliosis Study
Acronym: IV-KIDS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Association for the Advancement of Blood & Biotherapies (Unknown)
Responsible Party: Principal Investigator, Lisa Eisler, Assistant Professor of Anesthesiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAV9024
Record Dates: First submitted 2025-10-14; First posted 2025-10-20 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Scoliosis Correction; Iron Deficiency; Transfusion Blood; Surgery Complications; Spinal Fusion; Scoliosis Idiopathic Adolescent; Scoliosis Neuromuscular
Keywords: scoliosis; iron deficiency; blood transfusion; spinal fusion; iron supplementation
MeSH Terms: conditions — Iron Deficiencies; Scoliosis | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Intravenous ferric carboxymaltose (Experimental): Participants will receive ferric carboxymaltose, 15mg/kg up to 750mg intravenously, on the morning of surgery.
  Interventions: Drug: Ferric carboxymaltose IV
- Intravenous normal saline (Placebo Comparator): Patients will receive normal saline, intravenously, on the morning of surgery.
  Interventions: Drug: Normal Saline (Placebo)
- Observational follow-up (No Intervention): Participants who do not qualify for randomization may be invited to complete study measures through postoperative follow-up as part of an observational study.

INTERVENTIONS:
Drug: Ferric carboxymaltose IV — Ferric carboxymaltose is an intravenous treatment for iron deficiency.
  Arms: Intravenous ferric carboxymaltose
Drug: Normal Saline (Placebo) — Normal saline is the recommended diluent for ferric carboxymaltose, and on its own serves as the placebo control for this study.
  Arms: Intravenous normal saline

SUMMARY:
Adolescents and young adults undergoing spinal fusion surgery for the correction of scoliosis and other spinal deformity are at high risk of perioperative iron deficiency and anemia, yet the means and evidence for optimizing iron status have not been described in this setting. The proposed study is a randomized controlled trial of preoperative intravenous iron supplementation, to identify whether iron deficiency is a modifiable risk factor for adverse surgical outcomes such as red blood cell transfusion and diminished postoperative cognitive and physical capacity in this vulnerable population. Building evidence for patient blood management interventions such as iron supplementation is vital to ensuring high quality care of surgical patients and may reduce unnecessary transfusions amid recent blood shortages.

DETAILED DESCRIPTION:
Adolescents undergoing spinal fusion surgery for scoliosis and/or kyphosis are poised to benefit from preoperative iron supplementation. Spinal fusion carries a risk of large surgical blood losses and perioperative red blood cell transfusion, which are associated with adverse outcomes in this population. These patients are mostly adolescent females, a group more susceptible to iron deficiency and resulting anemia at baseline due to iron losses with menses, and who suffer an additional insult to iron stores during surgery. Nevertheless, iron status is not routinely monitored in this setting and there is no standard of care for preoperative iron supplementation. Iron is a nutritionally essential trace element important not only for red blood cell production, but also for muscle function and neurotransmitter synthesis and signaling. Therefore, supplementation of poor iron status is an important target for optimizing hemoglobin prior to surgery, reducing transfusion rates and associated complications such as alloimmunization, and improving patient outcomes. On its own and as the primary cause of anemia, iron deficiency was identified as the only risk factor for transfusion which is modifiable preoperatively. In addition, iron supplementation is shown to alleviate impairments of physical and cognitive capacity associated with even mild forms of iron deficiency in adolescent and young adult females. A pilot study conducted at Columbia University Irving Medical Center identified iron deficiency in 36% of scoliosis patients prior to surgery, with preoperative iron status highly correlated with iron status during surgical recovery. Consequently, the investigators plan to examine iron deficiency as a modifiable risk factor for transfusion and impaired postoperative cognitive and physical capacity in this vulnerable population. Previous trials of brief iron interventions in high-risk adult surgical patients, mostly with unknown iron status, do not inform the care of adolescents and were not designed to address postoperative functional outcomes. The investigators will therefore perform a single-center randomized controlled trial in which adolescents with scoliosis and/or kyphosis identified using physiologically-based serum markers of poor iron status will be randomized to a one time preoperative dose of IV ferric carboxymaltose or placebo, to test the hypotheses that preoperative iron supplementation 1) reduces the rate of red blood cell transfusion, 2) improves postoperative neurocognition compared to a preoperative baseline, and 3) improves patient reported physical functioning during recovery. This study aims to improve outcomes in this vulnerable population and provide evidence for patient blood management approaches to reduce transfusions amid recent severe blood shortages.

ELIGIBILITY:
Inclusion Criteria:

* 10 -19 years old
* diagnosis of scoliosis or kyphosis
* scheduled for imminent spinal fusion procedure (<6 weeks) at MS-CHONY
* Iron deficiency or hypoferritinemia, defined as serum ferritin less than or equal to 50 μg/L

Exclusion Criteria:

* C-reactive protein > 10 mg/L
* receiving nutritional support by report in the medical chart
* self-reported history of hypersensitivity reaction to iron-containing supplements
* self-reported history of receiving intravenous iron supplements
* self-reported history of iron overloaded state such as hereditary hemochromatosis or hemosiderosis
* objection to receiving red blood cell transfusions
* current pregnancy (identified by self-report or documentation of preoperative screening test in the medical record)
* prisoners
* patient or parent decides against study participation

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of perioperative RBC transfusion in iron deficient scoliosis patients undergoing spinal fusion | 4-30 days
  The patients that received a red blood cell transfusion either during procedure or postoperatively during their surgical hospitalization will be tallied.

SECONDARY OUTCOMES:
Percentage of Patients that experienced postoperative change in neurocognitive function | 2 to 3 months
  The Cognitive Battery of the NIH Toolbox is a brief, valid, and reliable instrument designed to provide outcome measures in epidemiologic and longitudinal research that can be used for comparisons across a wide range of studies and populations. Individual measure scores in the battery reflect Executive Function, Attention, Verbal and Nonverbal Memory, Language, Processing Speed, and Working Memory, yielding a composite score. This composite is scored on a T-score, with 100 representing the mean normalized by age and education level, and a standard deviation of 10. A score of 100 indicates performance that was at the national average for the test-taking participant's age. Scores of 85 or lower indicate below average cognitive function. A decline of function is measured by comparing the mean change from baseline in the Cognitive Function Composite Scores in the study groups.
Percentage of patients that experienced postoperative change in self-reported physical capacity | 2 to 3 months
  The PROMIS pediatric measures are a NIH Roadmap initiative to provide access to valid and reliable self-reported measures of health-related quality of life in children and adolescents. The PROMIS measures are scored on a T-score metric, where a score of 50 and standard deviation of 10 represents the average score for the general population in the United States. Higher PROMIS symptom scores indicate increased symptom burden, and higher PROMIS function scores indicate increased functioning. Decline would be identified through a mean change (decrease) from baseline in the Physical Functioning - Mobility scores; with secondary hypotheses for Physical Functioning - Upper Extremity, Physical Activity, and Fatigue.
Volume of perioperative RBC transfusion | 4 to 30 days
  The volume that each patient receives either during procedure or postoperatively during surgical hospitalization will be summed and average calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will make the determination to share or not share IPD at a later date.

REFERENCES:
- [Background] Qiu A, Fliginger D, Feit Y, Hassan F, Lenke LG, Li G, Hod EA, Eisler L. Estimating the prevalence of preoperative iron deficiency and its impact on red blood cell transfusion in adolescents undergoing scoliosis surgery: A pilot study. Transfusion. 2025 May;65(5):851-857. doi: 10.1111/trf.18246. Epub 2025 Apr 7. PMID 40191932